CLINICAL TRIAL: NCT05176353
Title: Implementation of a Diagnostic Stewardship Bundle for Ventilator-associated Pneumonia Among Mechanically-ventilated Patients
Brief Title: Ventilator-associated Pneumonia (VAP) Diagnostic Stewardship Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Owen Albin, Assistant Professor of Internal Medicine, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00203162; 5UL1TR002240-05 (NIH)
Record Dates: First submitted 2021-11-23; First posted 2022-01-04 (Actual); Results first posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: VAP - Ventilator Associated Pneumonia
Keywords: Antimicrobial stewardship; Ventilator-associated pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Intervention Model Description: Implementation of a VAP diagnostic stewardship bundled intervention targeting ordering, collection and reporting results of respiratory cultures among mechanically-ventilated patients. Interventions will be implemented through a custom order set within the institutional electronic medical record in 2-month sequential intervals. Safety, ICU-specific antibiotic utilization rates and adherence to study interventions will be monitored.
Masking Description: Due to the nature of this pilot trial the study will obtain an exemption from informed consent.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VAP diagnostic stewardship (Experimental): Intervention group - all patients hospitalized in study ICUs who were mechanically ventilated Feb 17 2022 - Feb 17 2023.
  Interventions: Other: VAP diagnostic stewardship bundle
- Pre-VAP diagnostic stewardship (No Intervention): Pre-intervention historical control group - all patients hospitalized in study ICUs who were mechanically ventilated Feb 17 2017-Feb 16 2022.
  While these patients were all mechanically ventilated, their treatment took place prior to the beginning of the study, under what standard or standards of care existed at the time. They received no treatment during the course of the study. No interventions could be assigned because their treatment was performed prior to study start date.

INTERVENTIONS:
Other: VAP diagnostic stewardship bundle — Multifaceted VAP diagnostic stewardship bundle targeting the respiratory culture testing workflow through a custom order set within the institutional electronic medical record. Interventions will be made at the three levels of the diagnostic testing pathway (ordering, collection and reporting of test results). Full details available in detailed study description.
  Arms: VAP diagnostic stewardship

SUMMARY:
This is a prospective pilot/feasibility trial of a bundled diagnostic stewardship intervention at the level of the microbiologic testing pathway in ventilator-associated pneumonia (VAP). The study utilized a pre/post design and was initially registered as a single-arm trial because the study intervention could only be applied prospectively to a single group (all patients hospitalized in study ICUs requiring ventilation during the trial intervention period). The study objectives are to safely and effectively reduce antibiotic overuse and its attendant hazards (adverse drug events, Clostridioides difficile diarrhea and generation of multidrug-resistant organisms) among mechanically-ventilated patients. Participating ICUs will have the following three modifications made in their respiratory culture workflows for mechanically-ventilated patients: 1) providers will be required to select a valid indication for respiratory culture performance (worsening ventilator requirements, purulent sputum production, and/or new radiographic infiltrate on chest imaging); 2) respiratory cultures will be preferentially obtained via bronchoscopic or nonbronchoscopic BAL (by respiratory therapists) rather than via endotracheal aspiration; and 3) BAL samples will be sent for cell count and differentials, and respiratory culture results will not be released for samples with <50% neutrophils. The study will carefully monitor adherence to study interventions, ICU-specific antibiotic utilization rates, and important safety metrics including rates of mortality, ventilator-dependence and ventilator-associated events.

The trial hypotheses are:

* Implementation of a VAP diagnostic stewardship bundle will be successfully implemented without significant increases in mortality or ventilator-associated events.
* Implementation of a VAP diagnostic stewardship bundle will be associated with a reduction in ICU-specific antibiotic utilization rates

DETAILED DESCRIPTION:
Overdiagnosis of ventilator-associated pneumonia (VAP) is common among mechanically-ventilated patients and contributes to antibiotic overuse and the generation of multidrug resistant organisms within intensive care units (ICUs). Identification of interventions that safely and effectively lower VAP overdiagnosis and antibiotic overuse are important for antimicrobial stewardship programs. Antibiotic stewardship interventions targeting VAP have heretofore focused on therapeutic interventions-antibiotic de-escalation or discontinuation-in established VAP cases, but have not leveraged interventions at the level of the VAP diagnostic testing pathway to minimize overdiagnosis in the first place. Current microbiologic testing practices-specifically, indiscriminate ordering, collection and interpretation of respiratory cultures-incents VAP overdiagnosis and antibiotic overuse.

This is a prospective pilot/feasibility trial of a bundled diagnostic stewardship intervention targeting the microbiologic diagnostic testing pathway among mechanically-ventilated patients. The study utilized a pre/post design and was initially registered as a single-arm trial because the study intervention could only be applied prospectively to a single group (all patients hospitalized in study ICUs requiring ventilation during the trial intervention period). This pilot/feasibility trial will implement system-based changes within ICUs in microbiologic diagnostic testing workflows with the goal of safely lowering antibiotic utilization rates in mechanically-ventilated patients. Specifically, the study will sequentially implement the following 3 changes in the diagnostic testing workflow for clinical providers:

1. Ordering respiratory cultures:

   1. Current workflow: respiratory cultures can be ordered by frontline clinical providers without preconditions.
   2. Study intervention: frontline clinical providers will be required to select a valid indication for respiratory culture collection through a custom order set in the institutional electronic medical record (EMR).
2. Collection of respiratory cultures:

   1. Current workflow: providers may collect endotracheal aspirates (proximal lung secretions) or bronchoalveolar lavage (distal lung secretions) for analysis.
   2. Study intervention: providers will be required to preferentially use only bronchoalveolar lavage (BAL) to minimize false positive test results (assuming no contraindications to BAL performance). This will be accomplished through a custom order set in the institutional EMR.
3. Reporting of respiratory cultures:

   1. Current workflow: positive respiratory culture results are automatically released in the EMR, regardless of likelihood of infection.
   2. Study intervention: respiratory culture results will be automatically released in the EMR only for BAL samples with a polymorphonuclear (PMN) percentage of >50% (to minimize false positive test results). Respiratory culture results for BAL samples with PMN% <50% will be released if the primary team calls the microbiology lab directly and requests result release.

All proposed interventions are within the standard of care for routine clinical practice, but have not been operationalized in parallel to each other and studied explicitly with the goal of reducing antibiotic overuse. The first two study interventions will be implemented at the beginning of the trial period and the final study intervention will be implemented 6 months after. The interventions will be operationalized through use of a custom order set in the institutional EMR and modifications to Clinical Microbiology Laboratory Workflows, as well as through bimonthly provider educational sessions performed by study personnel during morning ICU rounds. Use of the clinical decision support tool within the EMR by frontline providers will be entirely volitional.

The study population in this trial includes all patients admitted to participating study ICUs for routine clinical care. Providers will engage in routine clinical care utilizing the aforementioned modified diagnostic testing workflows and the study will compare safety outcomes and ICU antibiotic utilization rates pre- and post-intervention implementation.

Healthcare providers in participating ICUs will provide routine clinical care utilizing these novel diagnostic testing workflows. Adherence to study interventions by these healthcare providers will be assessed during this study to inform project feasibility on a larger scale.

ELIGIBILITY:
Inclusion Criteria Patients included:

* All patients hospitalized within the Michigan Medicine Cardiac Care Unit (CCU, 7D) and the Michigan Medicine Critical Care Medicine Unit (CCMU, 6D)

Exclusion Criteria Patients included:

* For the study intervention requiring performance of bronchoalveolar lavage rather than endotracheal aspirate for respiratory culture collection, the following are exclusion criteria for performance of bronchoalveolar lavage:

  * international normalized ratio (INR)>2,
  * platelet count <50,
  * gross blood in endotracheal secretions,
  * ratio of arterial oxygen partial pressure (PaO2 in mmHg) to fractional inspired oxygen (FiO2), ratio (P/F ratio)<80,
  * major lung surgery within prior 30 days.

Inclusion Criteria healthcare providers included:

* healthcare providers working in units (CCU and CCMU) as part of routine clinical care.

Exclusion Criteria healthcare providers included:

* healthcare providers that are not as part of routine care in CCU and CCMU

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4892 (Actual)
Dates: Start 2022-02-11 (Actual); Primary Completion 2023-02-12 (Actual); Study Completion 2023-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Owen Albin, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The entire study operated under waiver of consent. There was no "assignment" to the historical control arm. Rather, there was a collection of data retrospectively from persons on ventilators during the five-year period preceding the intervention period.
Groups:
- Pre-VAP Diagnostic Stewardship: Pre-intervention historical control group - all patients hospitalized in study ICUs who were mechanically ventilated Feb 17, 2017- Feb 16, 2022.
- VAP Diagnostic Stewardship: Intervention group - all patients hospitalized in study ICUs who were mechanically ventilated Feb 2022 - Feb 2023.
  VAP diagnostic stewardship bundle: Multifaceted VAP diagnostic stewardship bundle targeting the respiratory culture testing workflow through a custom order set within the institutional electronic medical record. Interventions will be made at the three levels of the diagnostic testing pathway (ordering, collection and reporting of test results). Full details available in detailed study description.
Period: Overall Study
Arm/Group | Pre-VAP Diagnostic Stewardship | VAP Diagnostic Stewardship
Started | 4205 | 687
Completed | 4205 | 687
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- VAP Diagnostic Stewardship: Intervention group - all patients hospitalized in study ICUs who were mechanically ventilated Feb 17, 2022 - Feb 17, 2023.
  VAP diagnostic stewardship bundle: Multifaceted VAP diagnostic stewardship bundle targeting the respiratory culture testing workflow through a custom order set within the institutional electronic medical record. Interventions will be made at the three levels of the diagnostic testing pathway (ordering, collection and reporting of test results). Full details available in detailed study description.
- Total: Total of all reporting groups
Arm/Group | Pre-VAP Diagnostic Stewardship | VAP Diagnostic Stewardship | Total
Number analyzed (Participants) | 4205 | 687 | 4892
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.7 (16.2) | 57.8 (16.8) | 58.6 (16.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1705 | 277 | 1982
  Male | 2500 | 410 | 2910
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 609 | 103 | 712
  White | 3303 | 517 | 3820
  Other | 293 | 67 | 360
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4205 | 687 | 4892

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Deaths in the Pre vs Post-intervention Time Periods Among Study Participants Per 1000 Mechanically Ventilated Patient Days
Description: The number of deaths that occur across the entire study population will be divided by every 1000 days that the total number of patients were hospitalized in study ICUs, receiving mechanical ventilation. Data was collected retrospectively for 5 years prior to the intervention and for 1 year during the intervention period.
Time Frame: During the period of mechanical ventilation (generally ranging between 1-2 days and 1 year).
Measure: Number (95% Confidence Interval); unit: Deaths per 1000 patient-days
Arm/Group | Pre-VAP Diagnostic Stewardship | VAP Diagnostic Stewardship
Number analyzed (Participants) | 4205 | 687
Deaths per 1000 patient-days | 72 [62 to 75] | 73 [64 to 82]
Statistical Analysis 1: Comparison: Pre-VAP Diagnostic Stewardship vs VAP Diagnostic Stewardship; Test type: Superiority; p = 0.86, Z-score test for person-time rates

2. Primary Outcome: Change in Ventilator-associated Events (V-A Events) (Using Centers for Disease Control/National Healthcare Safety Network Definitions) Per 1000 Patient Days
Description: The change in ventilator-associated events that occur across the entire study population will be divided by every 1000 days that the total number of patients were hospitalized in study ICUs, receiving mechanical ventilation, as shown by comparing pre-intervention data to post-intervention data. Data was collected retrospectively for 5 years prior to the intervention and for 1 year during the intervention period.
Time Frame: During the period of mechanical ventilation (generally ranging between 1-2 days and 1 year).
Measure: Number (95% Confidence Interval); unit: V-A events per 1000 pt days
Arm/Group | Pre-VAP Diagnostic Stewardship | VAP Diagnostic Stewardship
Number analyzed (Participants) | 4205 | 687
V-A events per 1000 pt days | 15 [13 to 17] | 10 [7 to 14]
Statistical Analysis 1: Comparison: Pre-VAP Diagnostic Stewardship vs VAP Diagnostic Stewardship; Test type: Superiority; p = 0.05, Z-score test for person-time rates

3. Primary Outcome: Median Duration of Mechanical Ventilation Per Patient
Time Frame: During the period of mechanical ventilation (generally ranging between 1-2 days and 1 year).
Measure: Median (Inter-Quartile Range); unit: Calendar Days
Groups:
- VAP Diagnostic Stewardship: Intervention group - all patients hospitalized in study ICUs who were mechanically ventilated Feb 17, 2022 - Feb 17,2023.
  VAP diagnostic stewardship bundle: Multifaceted VAP diagnostic stewardship bundle targeting the respiratory culture testing workflow through a custom order set within the institutional electronic medical record. Interventions will be made at the three levels of the diagnostic testing pathway (ordering, collection and reporting of test results). Full details available in detailed study description.
Arm/Group | Pre-VAP Diagnostic Stewardship | VAP Diagnostic Stewardship
Number analyzed (Participants) | 4205 | 687
Calendar Days | 3 [2 to 7] | 3 [2 to 7]
Statistical Analysis 1: Comparison: Pre-VAP Diagnostic Stewardship vs VAP Diagnostic Stewardship; Test type: Superiority; p = 0.59, Kruskal-Wallis

4. Secondary Outcome: Number of Positive Respiratory Cultures (RCs) Per 1,000 Mechanically-ventilated Patient Days (MVPDs)
Description: Positive respiratory cultures were defined as any respiratory culture growing a bacterial organism, regardless of total colony-forming units/mL
Time Frame: During the period of mechanical ventilation (generally ranging between 1-2 days and 1 year).
Measure: Number (95% Confidence Interval); unit: positive RCs per 1,000 MVPDs
Arm/Group | Pre-VAP Diagnostic Stewardship | VAP Diagnostic Stewardship
Number analyzed (Participants) | 4205 | 687
positive RCs per 1,000 MVPDs | 127 [122 to 131] | 102 [92 to 112]
Statistical Analysis 1: Comparison: Pre-VAP Diagnostic Stewardship vs VAP Diagnostic Stewardship; Test type: Superiority; p < 0.01, Z-score test for person-time rates

5. Secondary Outcome: Total ICU Antibiotic Utilization Rates
Description: Rates are shown as total antibiotic days of therapy per 1000 mechanically-ventilated patient days. A "Day of therapy" is defined as a calendar day in which a patient received a systemically-administered antibiotic, regardless of dose. Receipt of multiple, unique antibiotics on a given calendar day were counted cumulatively, that is, if a patient received 3 unique antibiotics that was counted as three days of therapy.
Time Frame: During the period of mechanical ventilation (generally ranging between 1-2 days and 1 year).
Measure: Number (95% Confidence Interval); unit: days of therapy per 1000 patient-days
Arm/Group | Pre-VAP Diagnostic Stewardship | VAP Diagnostic Stewardship
Number analyzed (Participants) | 4205 | 687
days of therapy per 1000 patient-days | 1361 [1346 to 1376] | 1335 [1300 to 1372]
Statistical Analysis 1: Comparison: Pre-VAP Diagnostic Stewardship vs VAP Diagnostic Stewardship; Test type: Superiority; p = 0.20, Z-score test for person-time rates

6. Secondary Outcome: Broad-spectrum ICU Antibiotic Utilization Rates
Description: Utilization rates are shown as broad-spectrum antibiotic days of therapy per 1000 mechanically-ventilated patient days. Broad-spectrum antibiotics were defined as antibiotics with expected coverage against methicillin-resistant Staphylococcus aureus or Pseudomonas aeruginosa. A "day of therapy" is defined as a calendar day in which a patient received a systemically-administered antibiotic, regardless of dose. Receipt of multiple, unique antibiotics on a given calendar day were counted cumulatively, that is, if a patient received 3 unique antibiotics that was counted as three days of therapy. .
Time Frame: During the period of mechanical ventilation (generally ranging between 1-2 days and 1 year).
Measure: Number (95% Confidence Interval); unit: days of therapy per 1000 patient-days
Groups:
- VAP Diagnostic Stewardship: Intervention group - all patients hospitalized in study ICUs who were mechanically ventilated Feb 17, 2022 - Feb 17, 2023. (ADD ACTUAL DATES)
  VAP diagnostic stewardship bundle: Multifaceted VAP diagnostic stewardship bundle targeting the respiratory culture testing workflow through a custom order set within the institutional electronic medical record. Interventions will be made at the three levels of the diagnostic testing pathway (ordering, collection and reporting of test results). Full details available in detailed study description.
Arm/Group | Pre-VAP Diagnostic Stewardship | VAP Diagnostic Stewardship
Number analyzed (Participants) | 4205 | 687
days of therapy per 1000 patient-days | 1199 [1177 to 1205] | 1149 [1116 to 1184]
Statistical Analysis 1: Comparison: Pre-VAP Diagnostic Stewardship vs VAP Diagnostic Stewardship; Test type: Superiority; p = 0.03, Z-score test for person-time rates

7. Secondary Outcome: Number of Respiratory Cultures Ordered Per 1000 Mechanically-ventilated Patient Days
Time Frame: During the period of mechanical ventilation (generally ranging between 1-2 days and 1 year).
Measure: Number (95% Confidence Interval); unit: Cultures ordered per 1000 patient-days
Arm/Group | Pre-VAP Diagnostic Stewardship | VAP Diagnostic Stewardship
Number analyzed (Participants) | 4205 | 687
Cultures ordered per 1000 patient-days | 334 [327 to 341] | 268 [252 to 285]
Statistical Analysis 1: Comparison: Pre-VAP Diagnostic Stewardship vs VAP Diagnostic Stewardship; Test type: Superiority; p < 0.01, Z-score test for person-time rates

8. Secondary Outcome: Percentage of Respiratory Cultures Obtained by Bronchoalveolar Lavage (BAL)
Time Frame: During the period of mechanical ventilation (generally ranging between 1-2 days and 1 year).
Population: Some providers ordered more than one culture per patient over the course of their hospital stay.
Measure: Number; unit: percentage of respiratory cultures
Units Other Than Participants: respiratory cultures obtained
Arm/Group | Pre-VAP Diagnostic Stewardship | VAP Diagnostic Stewardship
Number analyzed (Participants) | 4205 | 687
Number analyzed (respiratory cultures obtained) | 7753 | 1049
percentage of respiratory cultures | 53.1 | 56.9
Statistical Analysis 1: Comparison: Pre-VAP Diagnostic Stewardship vs VAP Diagnostic Stewardship; Test type: Superiority; p = .05, Chi-squared

9. Secondary Outcome: Percentage of Respiratory Cultures From BAL Samples With Alveolar Neutrophils <50% Following Study Intervention.
Time Frame: 6 months post-intervention
Population: This outcome measure only applied to the post-intervention arm. This was an optional test that providers could order, but many providers cancelled the test. Thus few BAL cell count/differentials were sent.
Measure: Number; unit: Percentage of respiratory cultures
Units Other Than Participants: tests
Arm/Group | VAP Diagnostic Stewardship
Number analyzed (Participants) | 16
Number analyzed (tests) | 22
Percentage of respiratory cultures | 4.3

ADVERSE EVENTS:
Time Frame: Up to 6 years (including 5 years pre-intervention and 1-year post intervention).
Description: Apart from in-hospital mortality, the only adverse event data collected was ventilator-associated events (VAEs). VAE numbers are complete and accurate, but number of unique persons affected by VAEs was not collected. Given the constraints of the clinicaltrials.gov reporting system, the number of events is replicated in number of persons affected. In fact, the number of persons affected could be equal to or less than that number. No non-serious AE data was collected, thus the denominator is 0.
Arm/Group | Pre-VAP Diagnostic Stewardship | VAP Diagnostic Stewardship
All-Cause Mortality (participants affected / at risk) | 1666/4205 | 284/687
Serious Adverse Events (participants affected / at risk) | 278/4205 | 34/687
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre-VAP Diagnostic Stewardship (N=4205) | VAP Diagnostic Stewardship (N=687)
ventilator associated events (Respiratory, thoracic and mediastinal disorders) | 278 (278) | 34 (34)

LIMITATIONS AND CAVEATS:
Ventilator-Associated Event numbers are complete and accurate, but number of unique persons affected by ventilator-associated events was not collected. Given the constraints of the clinicaltrials.gov reporting system, the number of events is replicated in number of persons affected. In fact, the number of persons affected could be equal to or less than that number.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-04): https://cdn.clinicaltrials.gov/large-docs/53/NCT05176353/Prot_SAP_000.pdf